CLINICAL TRIAL: NCT02328612
Title: Phase I, Randomized, Parallel Group, Placebo Control, Unicentric, Interventional Study to Assess the Effect of Expanded Human Allogeneic Adipose-derived Mesenchymal Adult Stem Cells on the Human Response to Lipopolysaccharyde in Human Volunteers
Brief Title: Randomized, Parallel Group, Placebo Control, Unicentric, Interventional Study to Assess the Effect of Expanded Human Allogeneic Adipose-derived Mesenchymal Adult Stem Cells on the Human Response to Lipopolysaccharyde in Human Volunteers
Acronym: CELLULA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Cellerix (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cx611-0102
Record Dates: First submitted 2014-12-11; First posted 2014-12-31 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- First arm (Experimental): 250,000 cells/kg will be administered via intravenous infusion.
  Interventions: Other: Intravenous infusion of cells
- Second arm (Experimental): 1,000,000 cells/kg will be administered via intravenous infusion.
  Interventions: Other: Intravenous infusion of cells
- Third arm (Experimental): 4,000,000 cells/kg will be administered via intravenous infusion.
  Interventions: Other: Intravenous infusion of cells
- Fourth arm (Placebo Comparator): Placebo (Ringer's lactate solution) volume according to subject's weight.
  Interventions: Other: Intravenous infusion of cells

INTERVENTIONS:
Other: Intravenous infusion of cells — The treatment administration will be infused intravenously to the subjects after randomization:
  An hour after the end of the eASCs administration, all subjects will be given an intravenous dose of LPS. Subjects will be allowed to leave in the evening once deemed clinically stable by the investigator.

SUMMARY:
Phase I, randomized, parallel group, placebo control, unicentric, interventional study. Thirty two healthy male volunteers aged between 18-35 years will be randomized into the eASCs or placebo group if they meet all the inclusion criteria at a 3:1 ratio.

The treatment administration will be infused intravenously to the following groups after randomization:

* First arm: 250,000 cells/kg
* Second arm: 1 million cells/kg
* Third arm: 4 million cells/kg
* Fourth arm: placebo according to their weight.

An hour after the end of the eASCs administration, all subjects will be given an intravenous dose of LPS. Subjects will be allowed to leave in the evening once deemed clinically stable by the investigator.

DETAILED DESCRIPTION:
Medicinal product Suspension of expanded adipose-derived allogeneic adult stem cells (eASCs) at a single dose of 250,000 cells/kg, 1 million cells/kg or 4 million cells/kg by intravenous infusion after suspension in Ringer's lactate solution.

Control Placebo (Ringer's lactate solution) Objectives To investigate the effect of eASCs on the inflammatory response to intravenous LPS in humans.

Design Phase I, randomized, parallel group, placebo control, unicentric, interventional study. Thirty two healthy male volunteers aged between 18-35 years will be randomized into the eASCs or placebo group if they meet all the inclusion criteria at a 3:1 ratio.

The treatment administration will be infused intravenously to the following groups after randomization:

* First arm: 250,000 cells/kg
* Second arm: 1 million cells/kg
* Third arm: 4 million cells/kg
* Fourth arm: placebo according to their weight.

An hour after the end of the eASCs administration, all subjects will be given an intravenous dose of LPS. Subjects will be allowed to leave in the evening once deemed clinically stable by the investigator.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Healthy, as determined by a responsible physician, based on a medical evaluation including medical history, physical examination and laboratory tests carried out within 28 days prior to administration of eASCs (if applicable) and LPS. A subject with a clinical abnormality or laboratory parameter outside the reference range may be included only if the investigator judges that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
2. Male aged between 18 and 35 years, inclusive at the time of signing the informed consent
3. Male subjects (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in activity in which conception is possible while on study medication and for at least 28 days after taking the last dose of study medication
4. Must understand and voluntarily sign an informed consent form prior to the conduct of any study related assessment/procedures. Capable of giving written informed consent and able to comply with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Subject has had a major illness in the past 3 months or any significant chronic medical illness that the investigator would deem unfavourable for enrolment, including inflammatory diseases
2. Subjects with a history of malignancy
3. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease
4. Subject uses tobacco products
5. Subject has a history, within 3 years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, THC, methamphetamine)
6. History of alcoholism and/or drinking more than 5 units of alcohol per day
7. Any clinically relevant abnormality noted on the 12-lead ECG as judged by the investigator or an average QTc > 450 msec
8. The subject has received an investigational product within three months prior to day 1 of the current study
9. Use of prescription or non-prescription drugs and herbal and dietary supplements within 6 months unless in the opinion of the investigator the medication will not interfere with the study procedures or compromise subject safety
10. Transfusion of blood or blood products within 6 months prior to the inclusion in the study.
11. Subject has difficultly in donating blood or accessibility of a vein in left or right arm.
12. Subject has donated more than 350 mL of blood in last 3 months
13. Body mass index >28 kg/m2
14. Presence of a severe bleeding or thrombotic disorder
15. History of known pulmonary embolism or known secondary anti-phospholipid syndrome
16. Subjects known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
17. Known allergies or hypersensitivity to antibiotics, HSA, DMEM, materials of bovine origin, and Ringer's Lactate Solution
18. Any other issue that, in the opinion of the investigator, could be harmful to the subject or compromise interpretation of the data.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory response as measured by laboratory measurements and functional assays of innate immunology | Change from baseline markers up to 10 hours after LPS injection
  To investigate the effect of eASCs on the inflammatory response to intravenous LPS in humans.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Perlee D, van Vught LA, Scicluna BP, Maag A, Lutter R, Kemper EM, van 't Veer C, Punchard MA, Gonzalez J, Richard MP, Dalemans W, Lombardo E, de Vos AF, van der Poll T. Intravenous Infusion of Human Adipose Mesenchymal Stem Cells Modifies the Host Response to Lipopolysaccharide in Humans: A Randomized, Single-Blind, Parallel Group, Placebo Controlled Trial. Stem Cells. 2018 Nov;36(11):1778-1788. doi: 10.1002/stem.2891. Epub 2018 Aug 20. PMID 30063804